CLINICAL TRIAL: NCT01958281
Title: A Phase 2b, Open-Label Study of 200 mg or 400 mg Sofosbuvir+RBV for 24 Weeks in Genotype 1 or 3 and Ledipasvir/Sofosbuvir (LDV/SOF) Fixed Dose Combination (FDC) Tablet for 12 Weeks in Genotype 1 or 4 HCV Infected Subjects With Renal Insufficiency
Brief Title: Sofosbuvir Plus Ribavirin, or Ledipasvir/Sofosbuvir in Adults With HCV Infection and Renal Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0154; 2013-002897-30 (EudraCT Number)
Record Dates: First submitted 2013-10-06; First posted 2013-10-09 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SOF 200 mg + RBV 200 mg (Cohort 1) (Experimental): Participants with genotype 1 or 3 HCV infection will receive SOF 200 mg (2 × 100 mg tablets) plus RBV once daily for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV
- SOF 400 mg + RBV 200 mg (Cohort 2) (Experimental): Participants with genotype 1 or 3 HCV infection will receive SOF 400 mg (4 × 100 mg tablets or 1 × 400 mg tablet) plus RBV once daily for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV
- LDV/SOF (Cohort 3) (Experimental): Participants with genotype 1 or 4 HCV infection will receive LDV/SOF once daily for 12 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: SOF — Tablet(s) administered orally once daily
  Other Names: Sovaldi®; GS-7977
  Arms: SOF 200 mg + RBV 200 mg (Cohort 1); SOF 400 mg + RBV 200 mg (Cohort 2)
Drug: RBV — 200 mg tablet administered orally once daily
  Arms: SOF 200 mg + RBV 200 mg (Cohort 1); SOF 400 mg + RBV 200 mg (Cohort 2)
Drug: LDV/SOF — 90/400 mg fixed-dose combination (FDC) tablet administered orally once daily
  Other Names: Harvoni®
  Arms: LDV/SOF (Cohort 3)

SUMMARY:
The primary objectives of this study are to evaluate the safety and efficacy of sofosbuvir (SOF) plus ribavirin (RBV) for 24 weeks and ledipasvir/sofosbuvir (LDV/SOF) for 12 weeks, and to evaluate the steady state pharmacokinetics (PK) of SOF and its metabolites and LDV in participants with genotype (GT) 1, 3, or 4 hepatitis C virus (HCV) infection who have chronic renal insufficiency (impaired kidney function).

ELIGIBILITY:
Key Inclusion Criteria:

* Cohorts 1 and 2: chronic genotype 1 or 3 HCV infection
* Cohort 3: chronic genotype 1 or 4 HCV infection
* HCV RNA ≥ 10^4 IU/mL at screening
* Screening labs within defined thresholds
* Cirrhosis determination at screening

Key Exclusion Criteria:

* Females who are pregnant or nursing or males who have a pregnant partner
* Prior null response to pegylated interferon (Peg-IFN)+RBV therapy (Cohorts 1 and 2) or for individuals with cirrhosis, prior treatment failure with IFN-based therapy not resulting from treatment intolerance (Cohort 3)
* Current of prior history of hepatic decompensation
* Infection with hepatitis B virus (HBV) or HIV
* History of clinically significant illness (including psychiatric or cardiac) or any other medical disorder that may interfere with individual's treatment and/or adherence to the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (10):
- United States (7):
  - San Francisco, California
  - Miami, Florida
  - Chicago, Illinois
  - Detroit, Michigan
  - Rochester, New York
  - San Antonio, Texas
  - Seattle, Washington
- New Zealand (2):
  - Grafton, Auckland
  - Christchurch
- San Juan, Puerto Rico

REFERENCES:
- [Background] Gane EJ, Robson RA, Bonacini M, Maliakkal B, Kirby B, Liu L, et al. Safety, Antiviral Efficacy, and Pharmacokinetics of Sofosbuvir in Patients With Severe Renal Impairment [Poster 966]. The 65th Annual meeting of the American Association for the Study of Liver Diseases: The Liver Meeting (AASLD); 2014 November 07-11; Boston, MA.
- [Background] Martin P, Gane E, Ortiz-Lasanta G, Liu L, Sajwani K, Kirby B, et al. Safety and Efficacy of Treatment With Daily Sofosbuvir 400 mg + Ribavirin 200 mg for 24 Weeks in Genotype 1 or 3 HCV-Infected Patients With Severe Renal Impairment [Poster 1128]. American Association for the Study of Liver Diseases (AASLD); 2015 November 13-17; San Francisco, CA.
- [Background] Lawitz E, Landis CS, Maliakkal BJ, Bonacini M, Ortiz-Lasanta G, Zhang J, et al. Safety and Efficacy of Treatment with Once- Daily Ledipasvir/Sofosbuvir (90/400 mg) for 12 Weeks in Genotype 1 HCV-Infected Patients with Severe Renal Impairment [Abstract 1587]. The Liver Meeting® 2017 - The 68th Annual Meeting of the American Association for the Study of Liver Diseases (AASLD); 2017 20-24 October; Washington, D. C.
- [Derived] Lawitz E, Landis CS, Flamm SL, Bonacini M, Ortiz-Lasanta G, Huang J, Zhang J, Kirby BJ, De-Oertel S, Hyland RH, Osinusi AO, Brainard DM, Robson R, Maliakkal BJ, Gordon SC, Gane EJ. Sofosbuvir plus ribavirin and sofosbuvir plus ledipasvir in patients with genotype 1 or 3 hepatitis C virus and severe renal impairment: a multicentre, phase 2b, non-randomised, open-label study. Lancet Gastroenterol Hepatol. 2020 Oct;5(10):918-926. doi: 10.1016/S2468-1253(19)30417-0. Epub 2020 Jun 10. PMID 32531259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and New Zealand. The first participant was screened on 07 October 2013. The last study visit occurred on 19 October 2017.
Pre-assignment Details: 32 participants were screened for Cohorts 1 and 2 and 33 participants were screened for Cohort 3.
Groups:
- SOF 200 mg + RBV 200 mg (Cohort 1): Sofosbuvir (SOF) 200 mg tablet once daily + ribavirin (RBV) 200 mg tablet once daily for 24 weeks
- SOF 400 mg + RBV 200 mg (Cohort 2): SOF 400 mg tablet once daily + RBV 200 mg tablet once daily for 24 weeks
- LDV/SOF (Cohort 3): Ledipasvir/sofosbuvir (LDV/SOF) 90/400 mg fixed-dose combination (FDC) tablet for 12 weeks
Period: Overall Study
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
Started | 10 | 10 | 18
Completed | 4 | 6 | 18
Not Completed | 6 | 4 | 0
Not completed — Lack of Efficacy | 5 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Withdrew Consent | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of study drug.
Groups:
- SOF 200 mg + RBV 200 mg (Cohort 1): SOF 200 mg tablet once daily + RBV 200 mg tablet once daily for 24 weeks
- LDV/SOF (Cohort 3): LDV/SOF 90/400 mg FDC tablet for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3) | Total
Number analyzed (Participants) | 10 | 10 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (6.5) | 58 (9.0) | 57 (7.5) | 58.9 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 12 | 18
  Male | 6 | 8 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 4 | 7
  Not Hispanic or Latino | 8 | 9 | 14 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 5 | 4 | 10 | 19
  White | 2 | 5 | 8 | 15
  Asian | 1 | 0 | 0 | 1
  Hawaiian or Pacific Islander | 0 | 1 | 0 | 1
  Other | 2 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 7 | 6 | 1 | 14
  United States | 3 | 4 | 17 | 24
HCV genotype [Count of Participants; unit: Participants]
  Genotype 1a | 7 | 6 | 14 | 27
  Genotype 1b | 2 | 2 | 4 | 8
  Genotype 3a | 1 | 2 | 0 | 3
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 2 | 5 | 1 | 8
    CT | 6 | 4 | 11 | 21
    TT | 2 | 1 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were enrolled and took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 10 | 10 | 18
percentage of participants | 40.0 [12.2 to 73.8] | 60.0 [26.2 to 87.8] | 100.0 [81.5 to 100.0]

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: Up to 24 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 10 | 10 | 18
percentage of participants | 100.0 | 90.0 | 72.2

3. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased by at least 1 toxicity grade from baseline at any time postbaseline up to the date of last dose of study drug plus 30 days.
Time Frame: Up to 24 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 10 | 10 | 18
percentage of participants | 100.0 | 100.0 | 100.0

4. Primary Outcome: Percentage of Participants Experiencing Clinically Significant 12-lead Electrocardiogram (ECG) Abnormalities
Time Frame: Up to 24 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 10 | 10 | 18
percentage of participants | 0 | 0 | 5.6

5. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events Associated With Vital Sign Abnormalities
Time Frame: Up to 24 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 10 | 10 | 18
percentage of participants | 10.0 | 0 | 0

6. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 2 (Cohorts 1 and 2)
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2
Population: Participants in the PK Analysis Set (all enrolled participants who took at least 1 dose of study drug and have at least 1 nonmissing postdose PK concentration value) from Cohorts 1 and 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
h*ng/mL
  SOF: number analyzed (Participants) | 8 | 10
  SOF | 1093.9 (703.03) | 1630.5 (851.33)
  GS-566500 | 2120.2 (837.51) | 4026.2 (1848.50)
  GS-331007 | 31859.4 (12621.62) | 51989.6 (29461.91)
  RBV | 22253.9 (6860.72) | 23595.5 (9636.77)

7. Primary Outcome: PK Parameter: AUCtau of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 12 (Cohorts 1 and 2)
Description: as for outcome 6
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 12
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 8
h*ng/mL
  SOF: number analyzed (Participants) | 9 | 8
  SOF | 1302.7 (652.18) | 1571.3 (944.71)
  GS-566500 | 2223.2 (877.20) | 3213.9 (1221.71)
  GS-331007 | 31078.3 (16745.94) | 46810.1 (25249.07)
  RBV: number analyzed (Participants) | 8 | 8
  RBV | 45341.9 (8712.71) | 50471.2 (23077.43)

8. Primary Outcome: PK Parameter: AUCtau of SOF, Its Metabolites (GS-566500 and GS-331007), and LDV at Week 2 or 4 (Cohort 3)
Description: as for outcome 6
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2 or 4
Population: Participants in the PK Analysis Set from Cohort 3 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 17
h*ng/mL
  SOF | 3536.8 (2040.59)
  GS-566500 | 7716.6 (3534.76)
  GS-331007 | 71463.3 (28979.92)
  LDV | 18460.1 (19999.95)

9. Primary Outcome: PK Parameter: Cmax of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 2 (Cohorts 1 and 2)
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
ng/mL
  SOF | 575.9 (487.66) | 976.8 (712.04)
  GS-566500 | 308.3 (132.60) | 538.3 (241.51)
  GS-331007 | 1750.0 (578.56) | 2721.4 (1452.86)
  RBV | 1373.1 (496.37) | 1373.8 (550.23)

10. Primary Outcome: PK Parameter: Cmax of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 12 (Cohorts 1 and 2)
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 12
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 8
ng/mL
  SOF | 903.9 (598.55) | 1422.9 (1390.47)
  GS-566500 | 352.2 (127.83) | 509.1 (216.71)
  GS-331007 | 1727.0 (775.37) | 2645.0 (1482.10)
  RBV: number analyzed (Participants) | 8 | 8
  RBV | 2458.8 (437.54) | 2589.4 (1159.66)

11. Primary Outcome: PK Parameter: Cmax of SOF, Its Metabolites (GS-566500 and GS-331007), and LDV at Week 2 or 4 (Cohort 3)
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2 or 4
Population: Participants in the PK Analysis Set from Cohort 3 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 17
ng/mL
  SOF | 2018.1 (1110.56)
  GS-566500 | 1021.6 (359.13)
  GS-331007 | 3570.0 (1325.31)
  LDV | 903.4 (844.70)

12. Primary Outcome: PK Parameter: Ctau of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 2 (Cohorts 1 and 2)
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
ng/mL
  SOF | NA (NA) — All values were below the limit of quantitation. | NA (NA) — All values were below the limit of quantitation.
  GS-566500 | 3.7 (7.88) | 20.8 (20.51)
  GS-331007 | 1023.0 (477.15) | 1736.1 (1110.41)
  RBV | 759.1 (240.04) | 818.8 (323.67)

13. Primary Outcome: PK Parameter: Ctau of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 12 (Cohorts 1 and 2)
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 12
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 9
ng/mL
  SOF | NA (NA) — All values were below the limit of quantitation. | NA (NA) — All values were below the limit of quantitation.
  GS-566500 | 2.3 (7.12) | 10.4 (11.07)
  GS-331007 | 952.5 (586.51) | 1356.0 (681.23)
  RBV | 1567.5 (529.35) | 1968.6 (884.99)

14. Primary Outcome: PK Parameter: Ctau of SOF, Its Metabolites (GS-566500 and GS-331007), and LDV at Week 2 or 4 (Cohort 3)
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2 or 4
Population: Participants in the PK Analysis Set from Cohort 3 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 16
ng/mL
  SOF | 2.9 (1.57)
  GS-566500 | 59.3 (88.08)
  GS-331007 | 2568.2 (1106.81)
  LDV | 705.0 (876.54)

15. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 10 | 10 | 18
percentage of participants | 40.0 [12.2 to 73.8] | 60.0 [26.2 to 87.8] | 100.0 [81.5 to 100.0]

16. Secondary Outcome: Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR4 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 10 | 10 | 18
percentage of participants | 40.0 [12.2 to 73.8] | 60.0 [26.2 to 87.8] | 100.0 [81.5 to 100.0]

17. Secondary Outcome: Percentage of Participants With Overall Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 10 | 10 | 18
percentage of participants | 50.0 | 40.0 | 0

18. Secondary Outcome: PK Parameter: AUClast of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 2 (Cohorts 1 and 2)
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
h*ng/mL
  SOF | 885.0 (710.72) | 1607.7 (854.70)
  GS-566500 | 1973.3 (851.52) | 3965.7 (1900.25)
  GS-331007 | 31859.4 (12621.62) | 51989.6 (29461.91)
  RBV | 22253.9 (6860.72) | 23595.5 (9636.77)

19. Secondary Outcome: PK Parameter: AUClast of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 12 (Cohorts 1 and 2)
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 12
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
h*ng/mL
  SOF: number analyzed (Participants) | 10 | 8
  SOF | 1177.7 (674.86) | 1548.1 (955.12)
  GS-566500: number analyzed (Participants) | 10 | 8
  GS-566500 | 1867.1 (839.39) | 3133.0 (1230.39)
  GS-331007: number analyzed (Participants) | 10 | 8
  GS-331007 | 31078.3 (16745.94) | 46810.1 (25249.07)
  RBV | 45341.9 (8712.71) | 50471.2 (23077.43)

20. Secondary Outcome: PK Parameter: AUClast of SOF, Its Metabolites (GS-566500 and GS-331007), and LDV at Week 2 or 4 (Cohort 3)
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2 or 4
Population: Participants in the PK Analysis Set from Cohort 3 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 17
h*ng/mL
  SOF | 3519.3 (2045.64)
  GS-566500 | 7657.6 (3555.57)
  GS-331007 | 69177.7 (31267.56)
  LDV | 18044.3 (20210.19)

21. Secondary Outcome: PK Parameter: Clast of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 2 (Cohorts 1 and 2)
Description: Clast is defined as the last observable concentration of drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
ng/mL
  SOF | 68.0 (100.22) | 21.3 (22.22)
  GS-566500 | 37.6 (18.84) | 35.8 (21.06)
  GS-331007 | 1023.0 (477.15) | 1736.1 (1110.41)
  RBV | 759.1 (240.04) | 818.8 (323.67)

22. Secondary Outcome: PK Parameter: Clast of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 12 (Cohorts 1 and 2)
Description: Clast is defined as the last observable concentration of drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 12
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 8
ng/mL
  SOF | 100.7 (158.83) | 22.7 (30.15)
  GS-566500 | 72.2 (80.16) | 32.1 (22.04)
  GS-331007 | 952.5 (586.51) | 1412.9 (705.06)
  RBV | 1741.3 (417.42) | 2040.9 (917.23)

23. Secondary Outcome: PK Parameter: Clast of SOF, Its Metabolites (GS-566500 and GS-331007), and LDV at Week 2 or 4 (Cohort 3)
Description: Clast is defined as the last observable concentration of drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2 or 4
Population: Participants in the PK Analysis Set from Cohort 3 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 17
ng/mL
  SOF | 56.3 (216.91)
  GS-566500 | 70.5 (97.14)
  GS-331007 | 2570.6 (1071.71)
  LDV | 700.6 (848.90)

24. Secondary Outcome: PK Parameter: Tmax of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 2 (Cohorts 1 and 2)
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
hours
  SOF | 1.00 [0.50 to 2.00] | 1.50 [1.00 to 2.13]
  GS-566500 | 2.17 [2.00 to 3.97] | 4.00 [2.00 to 4.00]
  GS-331007 | 4.00 [4.00 to 4.00] | 6.00 [4.00 to 6.00]
  RBV | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00]

25. Secondary Outcome: PK Parameter: Tmax of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 12 (Cohorts 1 and 2)
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 12
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 8
hours
  SOF | 1.04 [1.00 to 2.00] | 0.50 [0.50 to 1.50]
  GS-566500 | 2.17 [1.93 to 4.00] | 2.00 [1.50 to 4.00]
  GS-331007 | 5.11 [4.00 to 6.05] | 5.00 [4.00 to 6.00]
  RBV: number analyzed (Participants) | 8 | 8
  RBV | 2.00 [1.00 to 2.17] | 1.50 [1.00 to 3.00]

26. Secondary Outcome: PK Parameter: Tmax of SOF, Its Metabolites (GS-566500 and GS-331007), and LDV at Week 2 or 4 (Cohort 3)
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2 or 4
Population: Participants in the PK Analysis Set from Cohort 3 with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 17
hours
  SOF | 1.00 [0.50 to 1.10]
  GS-566500 | 2.00 [2.00 to 2.02]
  GS-331007 | 4.02 [4.00 to 6.02]
  LDV | 6.00 [4.00 to 8.00]

27. Secondary Outcome: PK Parameter: Tlast of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 2 (Cohorts 1 and 2)
Description: Tlast is defined as the time (observed time point) of Clast.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
hours
  SOF | 4.00 [3.92 to 4.13] | 6.00 [4.00 to 8.13]
  GS-566500 | 12.00 [11.97 to 12.00] | 24.00 [12.00 to 24.00]
  GS-331007 | 24.00 [24.00 to 24.00] | 24.00 [24.00 to 24.00]
  RBV | 24.00 [24.00 to 24.00] | 24.00 [24.00 to 24.00]

28. Secondary Outcome: PK Parameter: Tlast of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 12 (Cohorts 1 and 2)
Description: Tlast is defined as the time (observed time point) of Clast.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 12
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 8
hours
  SOF | 4.00 [2.33 to 4.00] | 4.03 [4.00 to 6.00]
  GS-566500 | 12.00 [10.00 to 12.02] | 24.00 [12.00 to 24.00]
  GS-331007 | 24.00 [24.00 to 24.00] | 24.00 [24.00 to 24.00]
  RBV: number analyzed (Participants) | 8 | 8
  RBV | 24.00 [24.00 to 24.00] | 24.00 [24.00 to 24.00]

29. Secondary Outcome: PK Parameter: Tlast of SOF, Its Metabolites (GS-566500 and GS-331007), and LDV at Week 2 or 4 (Cohort 3)
Description: Tlast is defined as the time (observed time point) of Clast.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2 or 4
Population: Participants in the PK Analysis Set from Cohort 3 with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 17
hours
  SOF | 12.00 [12.00 to 12.00]
  GS-566500 | 24.00 [24.00 to 24.00]
  GS-331007 | 24.00 [24.00 to 24.00]
  LDV | 24.00 [24.00 to 24.00]

30. Secondary Outcome: PK Parameter: λz of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 2 (Cohorts 1 and 2)
Description: λz is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 were analyzed.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
1/hour
  SOF | 1.0419 (0.28621) | 1.0155 (0.33118)
  GS-566500 | 0.2078 (0.04748) | 0.1771 (0.05802)
  GS-331007 | 0.0275 (0.01331) | 0.0273 (0.01711)
  RBV | 0.0165 (0.00524) | 0.0141 (0.00658)

31. Secondary Outcome: PK Parameter: λz of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 12 (Cohorts 1 and 2)
Description: as for outcome 30
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 12
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 8
1/hour
  SOF: number analyzed (Participants) | 9 | 8
  SOF | 1.4002 (0.29086) | 1.2154 (0.24100)
  GS-566500 | 0.2232 (0.05244) | 0.1818 (0.06121)
  GS-331007 | 0.0332 (0.01388) | 0.0313 (0.02100)
  RBV: number analyzed (Participants) | 8 | 8
  RBV | 0.0124 (0.00580) | 0.0085 (0.00509)

32. Secondary Outcome: PK Parameter: λz of SOF, Its Metabolites (GS-566500 and GS-331007), and LDV at Week 2 or 4 (Cohort 3)
Description: as for outcome 30
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2 or 4
Population: Participants in the PK Analysis Set from Cohort 3 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 16
1/hour
  SOF | 0.6033 (0.24057)
  GS-566500 | 0.1705 (0.04602)
  GS-331007 | 0.0214 (0.01222)
  LDV | 0.0305 (0.01226)

33. Secondary Outcome: PK Parameter: t1/2 of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 2 (Cohorts 1 and 2)
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 10
hours
  SOF: number analyzed (Participants) | 8 | 10
  SOF | 0.67 [0.59 to 0.75] | 0.67 [0.57 to 0.87]
  GS-566500 | 3.31 [2.95 to 3.98] | 3.88 [3.17 to 4.44]
  GS-331007 | 30.53 [19.14 to 43.25] | 29.05 [17.29 to 35.15]
  RBV | 46.89 [41.03 to 47.87] | 56.43 [43.06 to 71.53]

34. Secondary Outcome: PK Parameter: t1/2 of SOF, Its Metabolites (GS-566500 and GS-331007), and RBV at Week 12 (Cohorts 1 and 2)
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 12
Population: Participants in the PK Analysis Set from Cohorts 1 and 2 with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2)
Number analyzed (Participants) | 10 | 8
hours
  SOF: number analyzed (Participants) | 9 | 8
  SOF | 0.48 [0.45 to 0.49] | 0.57 [0.48 to 0.67]
  GS-566500 | 3.03 [2.72 to 3.96] | 3.88 [2.93 to 4.79]
  GS-331007 | 22.03 [18.76 to 27.96] | 33.54 [13.61 to 45.15]
  RBV: number analyzed (Participants) | 8 | 8
  RBV | 61.25 [45.37 to 88.73] | 91.62 [54.00 to 171.91]

35. Secondary Outcome: PK Parameter: t1/2 of SOF, Its Metabolites (GS-566500 and GS-331007), and LDV at Week 2 or 4 (Cohort 3)
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose at Week 2 or 4
Population: Participants in the PK Analysis Set from Cohort 3 with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | LDV/SOF (Cohort 3)
Number analyzed (Participants) | 16
hours
  SOF | 1.18 [1.11 to 1.47]
  GS-566500 | 4.02 [3.57 to 4.68]
  GS-331007 | 39.30 [30.38 to 54.89]
  LDV | 25.96 [18.25 to 31.89]

ADVERSE EVENTS:
Time Frame: Up to end of treatment (Week 12 or Week 24) plus 30 days
Description: Safety Analysis Set: participants who took at least 1 dose of study drug.
Arm/Group | SOF 200 mg + RBV 200 mg (Cohort 1) | SOF 400 mg + RBV 200 mg (Cohort 2) | LDV/SOF (Cohort 3)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/10 | 4/18
Other Adverse Events (participants affected / at risk) | 10/10 | 9/10 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF 200 mg + RBV 200 mg (Cohort 1) (N=10) | SOF 400 mg + RBV 200 mg (Cohort 2) (N=10) | LDV/SOF (Cohort 3) (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF 200 mg + RBV 200 mg (Cohort 1) (N=10) | SOF 400 mg + RBV 200 mg (Cohort 2) (N=10) | LDV/SOF (Cohort 3) (N=18)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Retching (Gastrointestinal disorders) | 0 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Chills (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 4
Peripheral swelling (General disorders) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Eczema infected (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1
Headache (Nervous system disorders) | 4 | 0 | 4
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 1
Irritability (Psychiatric disorders) | 2 | 0 | 0
Tearfulness (Psychiatric disorders) | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (7):
  • Study Protocol: Original (2013-07-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT01958281/Prot_000.pdf
  • Study Protocol: Amendment 1 (2013-09-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT01958281/Prot_001.pdf
  • Study Protocol: Amendment 2 (2014-02-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT01958281/Prot_002.pdf
  • Study Protocol: Amendment 3 (2015-02-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT01958281/Prot_003.pdf
  • Study Protocol: Amendment 4 (2015-04-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT01958281/Prot_004.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan for Cohorts 1 and 2 (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT01958281/SAP_005.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan for Cohort 3 (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT01958281/SAP_006.pdf